CLINICAL TRIAL: NCT07139613
Title: Evaluation of Zirconia Crown Restoring Endodontically Treated Posterior Teeth With Two Finish Line Designs and Two Occlusal Reduction Schemes(a Randomized Clinical Trial)
Brief Title: We Will Assess Zirconia Crown Restoring Endodontically Treated Posterior Teeth With Two Finish Line Designs and Two Occlusal Reduction Schemes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Saira Bibi, Registrar prosthodontics, Armed Forces Institute of Dentistry, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: zirconia crowns
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Zirconia Crowns
Keywords: Zirconia crowns assessment with two finish line design and two occlusal reduction schemes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (PS) (Active Comparator)
  Interventions: Other: Control group(PS)Planer occlusal scheme with rounded shoulder finish line
- First intervention group (FF)flat occlusal scheme with feather-edge finish line (Experimental): In this intervention group flat occlusal scheme and feather edge finish line design is followed
  Interventions: Procedure: First intervention group(FF) flat occlusal scheme with feather edge finish line
- Second intervention group (FS)flat occlusal scheme with rounded shoulder finish line (Experimental)
  Interventions: Procedure: Second intervention group(FS) flat occlusal with rounded shoulder finish line design

INTERVENTIONS:
Other: Control group(PS)Planer occlusal scheme with rounded shoulder finish line — Control group (PS) will have planer occlusal scheme with rounded shoulder finish line.
  Arms: Control group (PS)
Procedure: First intervention group(FF) flat occlusal scheme with feather edge finish line — First intervention group we will have flat occlusal scheme with feather edge finish line
  Arms: First intervention group (FF)flat occlusal scheme with feather-edge finish line
Procedure: Second intervention group(FS) flat occlusal with rounded shoulder finish line design — Second intervention will have flat occlusal scheme with rounded shoulder finish line design
  Arms: Second intervention group (FS)flat occlusal scheme with rounded shoulder finish line

SUMMARY:
Endodontically treated posterior teeth will be restored with zirconia crowns with two finish line designs(feather edge and rounded shoulder) and two occlusal reduction schemes(flat and planer).The crowns were designed with exocad software program .After cementation clinical performance in terms of marginal adaptation ,marginal discoloration, fracture and secondary caries was evaluated at 3 subsequent follow-up visits every 3months for 1 year.

DETAILED DESCRIPTION:
Endodontically treated posterior teeth require full coverage coronal restoration, as they are more prone to fracture as compared to vital teeth .Over past two decades restorative dentistry there has been a paradigm shift in restorative dentistry towards monolithic zirconia crowns because of its superior esthetics ,excellent biocompatibility ,and continually improving biomechanical properties. For the long term clinical success of zirconia crowns tooth preparation designs particularly finish line designs and occlusal reduction play significant role. Different finish lines designs such as chamfer and shoulder, play a role in marginal fit of restoration .While assessing zirconia crowns of two finish line designs and two occlusal reduction schemes the participants were divided into three groups based on preparation design: the control group PS (planer occlusal and rounded shoulder) ; first interventional group (flat occlusal and feather); Second interventional group (flat occlusal and rounded shoulder) .To minimize bias the outcome assessor ,participants and statistician were blinded and only investigator will not blinded. After cementation on subsequent follow-up of one year with every three months interval United states Public Health Services Criteria (USPHS) is used for marginal adaptation ,discoloration, fracture and secondary caries, and gingival index score system is used for gingival response.

Second interventional group FS (Flat occlusal + rounded shoulder)

ELIGIBILITY:
Inclusion Criteria:

* patients from both genders.
* age range 18-65 years.
* patients with endodontically treated posterior teeth.

Exclusion Criteria:

* vital teeth
* anterior teeth.
* edentulous patient.
* patient with history of significant systemic diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Gingival index score system and United States Public Health Services Criteria(USPHS) | One year
  Marginal adaptation ,marginal discoloration ,fracture and secondary caries evaluated using (USPHS) United States Public Health Services Criteria and gingival index score system is used to evaluate gingival response.

CONTACTS AND LOCATIONS:
Locations (1):
- Armed Forces Institute of Dentistry, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No